CLINICAL TRIAL: NCT03842046
Title: Comparison of Continuous Infusion of Noradrenaline Versus Phenylephrine During Cesarean Section Under Spinal Anesthesia. A Randomized Controlled Trial
Brief Title: Prevention of Hypotension During Cesarean Section
Acronym: NOR-PHEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Collaborators: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-PHEN
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hypotension Symptomatic; Obstetric Anesthesia Problems; Cesarean Section Complications; Vasoconstriction
Keywords: hypotension; phenylephrine; noradrenaline; cardiac output; fetal; maternal hemodynamics; cesarean section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine infusion (Active Comparator): phenylephrine infusion (30 mL/h corresponding to 50 μg/min)
  Interventions: Procedure: phenylephrine infusion
- norepinephrine infusion (Active Comparator): norepinephrine infusion (30 mL/h corresponding to 4 μg/min)
  Interventions: Procedure: norepinephrine infusion

INTERVENTIONS:
Procedure: phenylephrine infusion — In parturients allocated to the phenylephrine group, a phenylephrine infusion will be initiated as soon as spinal anesthesia is established
  Arms: phenylephrine infusion
Procedure: norepinephrine infusion — In parturients allocated to the norepinephrine group group, a phenylephrine infusion will be initiated as soon as spinal anesthesia is established
  Arms: norepinephrine infusion

SUMMARY:
The aim of this double-blind randomized study will be to compare a fixed-rate prophylactic noradrenaline infusion to a fixed-rate prophylactic phenylephrine infusion during elective cesarean section under combined spinal-epidural anesthesia

DETAILED DESCRIPTION:
* Spinal anesthesia is the anesthetic technique of choice for elective cesarean section.
* Spinal anesthesia can be complicated by hypotension, with incidence exceeding 80% occasionally. Hypotension can lead to nausea, emesis and a subjective feeling of discomfort due to cerebral hypoperfusion. If left untreated, severe or sustained hypotension can lead to decreased uteroplacental flow and fetal distress of premature or compromised fetuses while severe complications to the parturient might ensue, such as loss of consciousness, aspiration, apnea or cardiac arrest
* One of the standard techniques to avoid maternal hypotension is the administration of a continuous phenylephrine infusion while studies have demonstrated its superiority as compared to rescue bolus phenylephrine administration. Additionally, as compared to ephedrine, phenylephrine is associated with less neonatal acidosis and better maintenance of uteroplacental blood flow. However, phenylephrine can lead to baroreceptor-mediated reflex bradycardia, with untoward consequences for maternal cardiac output.
* Recently, noradrenaline has been shown to be effective in maintaining blood pressure in obstetric patients. Noradrenaline is a strong-alpha agonist with weak beta-action, too. Therefore, it might prove superior in maintaining cardiac output as compared to phenylephrine. There have been a few studies examining the use of noradrenaline as a continuous infusion in this context but the optimal dose and safety and efficacy profile of noradrenaline continuous infusion in obstetrics is yet to be determined
* In all parturients, standard hemodynamic monitoring will be applied. Baseline systolic arterial pressure will be considered the average of three consecutive measurements that will not differ more than 10% among them. All parturients will have a peripheral intravenous catheter placed in the upper extremity after baseline hemodynamic measurements are recorded and will be infused 5 mL/kg of hydroxyethylstarch (pre-loading) before the regional procedure.
* Study group allocation will taker place according to a computer-generated sequence of random numbers. A standard spinal anesthetic consisting of ropivacaine 0.75% 1.8 mL plus fentanyl 10 μg will be administered in the left lateraL position at the L3-4 or L4-5 vertebral interspace. The study infusion medication (either phenylephrine or norepinephrine, depending on group allocation) will be started at the same time cerebrospinal fluid is obtained, immediately before injection of spinal medications. After the intrathecal injection, patients will placed in the supine position with a left lateral tilt of the table to provide left uterine displacement and to prevent aortocaval compression. The spinal sensory level will be tested bilaterally by pinprick to ensure a T4 dermatomal level before surgical incision.
* Hemodynamic parameters (systolic arterial blood pressure, diastolic arterial blood pressure, mean arterial blood pressure and heart rate) will be measured and recorded at discrete timepoints throughout the operation (baseline, start of vasoactive agent administration, parturient at supine position, sympathetic block at T4, knife-to-skin, neonatal delivery, start of oxytocin administration, start of skin closure, end of operation.
* During the operation, a rescue dose of phenylephrine 50 μg will be administered when systolic arterial pressure drops below 80% of baseline in combination with heart rate>80 bpm. Ephedrine 5 mg will be administered when there is hypotension (systolic arterial pressure <80% of baseline) in combination with heart rate less than 80 bpm. Hypertensive episodes (systolic blood pressure >120% of baseline) will be treated with halving the infusion while when systolic arterial pressure increases above 130% of baseline the infusion will be discontinued and will be restarted when systolic blood pressure decreases below the upper limit of the target range (120% of baseline value).

ELIGIBILITY:
Inclusion Criteria:

* adult parturients, American Society of Anesthesiologists (ASA) I-II, singleton gestation>37 weeks
* elective cesarean section

Exclusion Criteria:

* Body Mass Index (BMI) >40 kg/m2
* Body weight <50 kg
* Body weight>100 kg
* height<150 cm
* height>180 cm
* multiple gestation
* fetal abnormality
* fetal distress
* active labor
* cardiac disease
* pregnancy-induced hypertension
* thrombocytopenia
* coagulation abnormalities
* use of antihypertensive medication during pregnancy
* communication or language barriers
* lack of informed consent
* contraindication for regional anesthesia

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
incidence of bradycardia | intraoperative
  any incidence of heart rate<60/min will be recorded

SECONDARY OUTCOMES:
need for vasoconstrictor | intraoperative
  parturient needed or not vasoconstrictor during the operation
type of vasoconstrictor administered | intraoperative
  phenylephrine verus ephedrine
number of bolus doses of vasoconstrictor administered | intraoperative
  number of provided interventions to maintain systolic blood pressure within the set limits will be recorded
total dose of vasoconstrictor administered | intraoperative
  total dose in mg for ephedrine or μg for phenylephrine
incidence of hypotension | intraoperative
  any occurrence of hypotension throughout the operation will be recorded (systolic arterial pressure<80% of baseline throughout the operation)
incidence of hypertension | intraoperative
  any incidence of systolic blood pressure >120% of baseline will be recorded
incidence of nausea/vomiting | intraoperative
  incidence of nausea and vomiting throughout the operation
neonatal Apgar score at 1 min | 1 min post delivery
  neonatal Apgar score will be recorded at 1 min after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
neonatal Apgar score at 5 min | 5 min post delivery
  neonatal Apgar score will be recorded at 5 min after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
neonatal blood gases | 1 min post delivery
  fetal cord blood analysis will be performed immediately post-delivery
glucose in neonatal blood | 1 min post delivery
  glucose will be measured in the cord blood gas sample taken immediately post-delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, Principal Investigator — Aretaieion University Hospital; Emmanouil Stamatakis, PhD, Principal Investigator — Alexandra General Hospital of Athens; Dimitrios Valsamidis, PhD, Principal Investigator — Alexandra General Hospital of Athens; Sofia Chatzilia, PhD, Principal Investigator — Alexandra General Hospital of Athens
Locations (2):
- Greece (2):
  - Aretaieion University Hospital, Athens
  - Alexandra General Hospital of Athens, Athens

REFERENCES:
- [Background] Afolabi BB, Lesi FE. Regional versus general anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004350. doi: 10.1002/14651858.CD004350.pub3. PMID 23076903
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Maayan-Metzger A, Schushan-Eisen I, Todris L, Etchin A, Kuint J. Maternal hypotension during elective cesarean section and short-term neonatal outcome. Am J Obstet Gynecol. 2010 Jan;202(1):56.e1-5. doi: 10.1016/j.ajog.2009.07.012. Epub 2009 Aug 28. PMID 19716536
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Background] Laudenbach V, Mercier FJ, Roze JC, Larroque B, Ancel PY, Kaminski M, Breart G, Diemunsch P, Subtil D, Lejus C, Fresson J, Arnaud C, Rachet B, Burguet A, Cambonie G; Epipage Study Group. Anaesthesia mode for caesarean section and mortality in very preterm infants: an epidemiologic study in the EPIPAGE cohort. Int J Obstet Anesth. 2009 Apr;18(2):142-9. doi: 10.1016/j.ijoa.2008.11.005. Epub 2009 Feb 4. PMID 19195873
- [Background] Ngan Kee WD, Khaw KS, Ng FF, Lee BB. Prophylactic phenylephrine infusion for preventing hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2004 Mar;98(3):815-21, table of contents. doi: 10.1213/01.ane.0000099782.78002.30. PMID 14980943
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Comparison of phenylephrine infusion regimens for maintaining maternal blood pressure during spinal anaesthesia for Caesarean section. Br J Anaesth. 2004 Apr;92(4):469-74. doi: 10.1093/bja/aeh088. Epub 2004 Feb 20. PMID 14977792
- [Background] Siddik-Sayyid SM, Taha SK, Kanazi GE, Aouad MT. A randomized controlled trial of variable rate phenylephrine infusion with rescue phenylephrine boluses versus rescue boluses alone on physician interventions during spinal anesthesia for elective cesarean delivery. Anesth Analg. 2014 Mar;118(3):611-8. doi: 10.1213/01.ane.0000437731.60260.ce. PMID 24299932
- [Background] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Background] Ngan Kee WD, Khaw KS, Lau TK, Ng FF, Chui K, Ng KL. Randomised double-blinded comparison of phenylephrine vs ephedrine for maintaining blood pressure during spinal anaesthesia for non-elective Caesarean section*. Anaesthesia. 2008 Dec;63(12):1319-26. doi: 10.1111/j.1365-2044.2008.05635.x. PMID 19032300
- [Background] Cooper DW, Carpenter M, Mowbray P, Desira WR, Ryall DM, Kokri MS. Fetal and maternal effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2002 Dec;97(6):1582-90. doi: 10.1097/00000542-200212000-00034. PMID 12459688
- [Background] Stewart A, Fernando R, McDonald S, Hignett R, Jones T, Columb M. The dose-dependent effects of phenylephrine for elective cesarean delivery under spinal anesthesia. Anesth Analg. 2010 Nov;111(5):1230-7. doi: 10.1213/ANE.0b013e3181f2eae1. Epub 2010 Sep 14. PMID 20841418
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435